CLINICAL TRIAL: NCT04923698
Title: Yoga on Postpartum Depression
Brief Title: Effect of Yoga on Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo Un110
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Yoga
Keywords: Yoga; Postpartum; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Group A (Control group): It consisted of 20 women and treated by antidepressant drugs only for 12 weeks. Group B (Study group): It consisted of 20 women and treated by the same antidepressant drugs as in group A and yoga program, 50 minutes daily,7 days per week for 12 weeks (Total 84 sessions).
Who Masked: Outcomes Assessor
Masking Description: using closed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga (Active Comparator): The yoga program consisted of 12 exercises, , 50 minutes daily, 7 days per week for 12 weeks (Total 84 sessions).
  Interventions: Other: yoga training
- antidepressant (Active Comparator): All women in group A were treated by antidepressant only for 12 weeks
  Interventions: Other: yoga training

INTERVENTIONS:
Other: yoga training — All women in group B were treated by the same antidepressant drugs as in group A and yoga program, 50 minutes daily, 7 days per week for 12 weeks (Total 84 sessions).

SUMMARY:
This study was conducted to investigate the effect of yoga on postpartum depression. Subjects: Forty primipara women with postpartum depression (PPD) selected randomly from Kasr El Ainy University Hospital in Cairo complaining of postpartum depression at least one month after childbirth shared in this study.

DETAILED DESCRIPTION:
This study was conducted to investigate the effect of yoga on postpartum depression. Subjects: Forty primipara women with postpartum depression (PPD) selected randomly from Kasr El Ainy University Hospital in Cairo complaining of postpartum depression at least one month after childbirth shared in this study. Group A (Control group): It consisted of 20 women and treated by antidepressant drugs only for 12 weeks. Group B (Study group): It consisted of 20 women and treated by the same antidepressant drugs as in group A and yoga program, 50 minutes daily,7 days per week for 12 weeks (Total 84 sessions).

ELIGIBILITY:
Inclusion Criteria:

* Their ages were ranged from 20-35 years
* Their body mass index was less than 30 kg/m2

Exclusion Criteria:

* cardiac arrhythmia,
* respiratory problems,
* uncontrolled Type I diabetes

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
BMI assessment | three months
  The weight and height of each woman in both groups (A & B) were measured

SECONDARY OUTCOMES:
Zung self-rating depression scale | three months
  There are ten positively worded and ten negatively worded questions. Each question is scored on a scale of 1 through 4

CONTACTS AND LOCATIONS:
Locations (1):
- Ghada Ebrahim Elrefaye, Giza, Egypt